CLINICAL TRIAL: NCT06159387
Title: "Randomized Double-blind Placebo-controlled Clinical Trial to Evaluate the Safety and Efficacy of the Use of Cannabis Sativa Extract in the Treatment of Cocaine and Crack Addicts."
Brief Title: Randomized, Double-blind, Placebo-controlled Cannabis Extract x Placebo for Cocaine Addicts
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, André Malbergier, MD, MPH, PhD, Head of Alcohol and Drugs Service, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 69721222.0.0000.0068
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Cocaine Dependence
Keywords: Crack/cocaine; Clinical trial; Cannabis extract; Pharmacotherapy
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: After admission, 60 patients are randomly allocated into 2 groups. A simple randomization are carried out in which the computer program generates a number (0 or 1) for each subject who enters the research. Zero is the the placebo group and 1 is the active drug group. Neither the evaluators nor the patients know which medication each research subject is taking. The laboratory provides identical solutions of active drug and placebo to ensure blinding of the research and only professionals in that laboratory know which is placebo or active drug.
Who Masked: Participant, Care Provider, Investigator
Masking Description: A simple randomization are carried out in which the computer program generates a number (0 or 1) for each subject who enters the research. Zero is the the placebo group and 1 is the active drug group. Neither the evaluators nor the patients know which medication each research subject is taking. The laboratory provides identical solutions of active drug and placebo to ensure blinding of the research and only professionals in that laboratory know which is placebo or active drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabis extract (Experimental): Thirty patients will receive cannabis extract (total daily dose) 384 mg of CBD and 11.4 mg of THC divided into one intake in the morning (1 mL of oily solution - 192 mg of CBD and 5.7 mg of THC) and one intake in the evening ( 1 mL of oily solution - 192 mg of CBD and 5.7 mg of THC) during breakfast and dinner and psychotherapy.
  Interventions: Drug: Cannabis Extract Oil SR Capsule
- Placebo (Placebo Comparator): The other 30 subjects will receive placebo (same volumes of oily solution without active ingredient) and psychotherapy. Titration will be done with an initial dose of 1 mL taken at night and increased over 2 days to 1 mL morning and night. Patients using placebo will make similar increments to maintain the blind nature of the study.
  Interventions: Drug: Cannabis Extract Oil SR Capsule

INTERVENTIONS:
Drug: Cannabis Extract Oil SR Capsule — After randomization, in a double blind model, subjects receive cannabis extract or placebo conditioned in identical vials with the same volume of substance.
  Everyone will undergo psychotherapy in the CBT (cognitive behavioral therapy) model

SUMMARY:
2.1. General To evaluate the efficacy and safety of a Cannabis sativa extract (CBD (Cannabidiol) + up to 0.3% THC (Delta-9-tetrahydrocannabinol)), compared to placebo, in the treatment of cocaine/crack use disorder.

2.2. Specifics

* Compare the amount and frequency of cocaine use between the group treated with Cannabis sativa extract and the placebo group
* Compare adherence to treatment between the group treated with Cannabis sativa extract and the placebo group
* Evaluate the prevalence and intensity of depressive and anxious symptoms in patients using Cannabis sativa extract compared to patients using placebo
* Evaluate the incidence and severity of side effects in the active group compared to placebo.

DETAILED DESCRIPTION:
The project is being developed at the Interdisciplinary Group for Alcohol and Drug Studies (GREA). GREA is a service of the Perdizes Institute - Department of Psychiatry of the Hospital das Clínicas of Medical School of the University of São Paulo that offers specialized treatment for addiction..

After admission, 60 crack/cocaine dependent patients are randomly allocated into 2 groups.

Neither the evaluators nor the patients know which medication each research subject is taking. The laboratory provides the medication and placebo in identical solutions to ensure blinding of the research.

Thirty patients receive (total daily dose) 384 mg of CBD and 11.4 mg of THC divided into one intake in the morning (1 mL of oily solution - 192 mg of CBD and 5.7 mg of THC) and one intake in the evening ( 1 mL of oily solution - 192 mg of CBD and 5.7 mg of THC) during breakfast and dinner and psychotherapy. The other 30 subjects receive placebo (same volumes of oily solution without active ingredient) and psychotherapy.

Titration will be done with an initial dose of 1 mL taken at night and increased over 2 days to 1 mL morning and night. Patients using placebo make similar increments to maintain the blind nature of the study.

Pharmacological treatments for other psychiatric disorders or clinical pathologies are maintained.

Psychotherapeutic treatment consists of weekly group cognitive behavioral therapy for 12 weeks for all patients and under the coordination of a psychologist trained in the field. Each session have a discussion topic. The groups have a maximum of 10 patients and, as this number is reached, a new group is started.

At admission, patients are assessed by the following questionnaires:

Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders (SCID5), Addiction Severity Index 6 (ASI 6), Patient Health Questionnaire-9 (PHQ-9), GAD-7 (General Anxiety Disorder-7), Timeline followback (TLFB), Minnesota Cocaine Craving Scale (MCCS).

Also at admission, patients are evaluated by the following blood tests:

Complete blood count, AST (aspartate aminotransferase), ALT (alanine aminotransferase), GGT (gamma-glutamyltransferase), Alkaline phosphatase, Amylase,Lipase, Fasting blood glucose, Beta-HCG (human chorionic gonadotropin), Total bilirubin and fractions, Urea, Creatinine, Sodium, Potassium, Coagulogram (PT and APTT), Anti-HIV, Ag HBS, Anti HBs, Serology for Syphilis, Serology for Hepatitis C. Those exams will be repeated 2 times throughout the research project.

Patients are assessed biweekly by physicians by the following questionnaires:

TLFB MCCS UKU (Udvalg for Kliniske Undersøgelser) scale for assessing side effects

Urine toxicology tests will be carried out in every physician assessment (biweekly)

Patients are treated for 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old Patients who meet the DSM-5 criteria for Cocaine use disorder.

Exclusion Criteria:

* Patients diagnosed with Schizophrenia and Bipolar Affective Disorder Patients with a history of severe head trauma Patients who used marijuana in the last month Patients who meet the criteria for other substances dependence besides crack/cocaine and tobacco.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-10-23 (Estimated); Study Completion 2025-10-23 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the extract of cannabis compared to placebo | biweekly
  The primary outcome will be the comparison of treatment efficacy between the active and placebo groups at weeks 1, 2, 4, 6, 8, 10 and 12. This outcome will be assessed through:
  Self-report of improvement by TLFB: The number of days of use and the amount of drugs consumed on those days are registered.
  Decrease in crack intensity measured by the MCCS instrument. The MCCS reports the frequency, intensity, and duration of the craving during the last week.
  Negative test for cocaine/crack by urine test indicates no use

SECONDARY OUTCOMES:
Safety of the extract of cannabis in patients with crack/cocaine use disorders admitted to treatment | biweekly
  Side effects are measured by UKU scale

CONTACTS AND LOCATIONS:
Overall Officials: Andre Malbergier, MD, MPH, PhD, Principal Investigator — Department of Psychiatry - University of São Paulo
Locations (1):
- Instituto Perdizes, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, ICF
Time Frame: October 2024 to october 2025
Access Criteria: Researchers in the field

REFERENCES:
- [Background] Karimi-Haghighi S, Razavi Y, Iezzi D, Scheyer AF, Manzoni O, Haghparast A. Cannabidiol and substance use disorder: Dream or reality. Neuropharmacology. 2022 Apr 1;207:108948. doi: 10.1016/j.neuropharm.2022.108948. Epub 2022 Jan 13. PMID 35032495
- [Background] Ledesma JC, Manzanedo C, Aguilar MA. Cannabidiol prevents several of the behavioral alterations related to cocaine addiction in mice. Prog Neuropsychopharmacol Biol Psychiatry. 2021 Dec 20;111:110390. doi: 10.1016/j.pnpbp.2021.110390. Epub 2021 Jun 19. PMID 34157334
- [Background] Mongeau-Perusse V, Brissette S, Bruneau J, Conrod P, Dubreucq S, Gazil G, Stip E, Jutras-Aswad D. Cannabidiol as a treatment for craving and relapse in individuals with cocaine use disorder: a randomized placebo-controlled trial. Addiction. 2021 Sep;116(9):2431-2442. doi: 10.1111/add.15417. Epub 2021 Feb 9. PMID 33464660